CLINICAL TRIAL: NCT06645340
Title: Does Nicotine Influence the Risk of Preeclampsia? A Prospective Study
Brief Title: Does Nicotine Influence the Risk of Preeclampsia?
Acronym: PRE_Smoking
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: EK-Nr.: 31-541 ES 18/19
Record Dates: First submitted 2024-10-15; First posted 2024-10-16 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Preeclampsia (PE); Endothelial Dysfunction; Hypertension in Pregnancy
Keywords: Preeclampsia Risk; Smoking; Endothelial Function; Arterial Stiffness; Retinal Microvasculature
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced; Smoking | interventions — Vascular Stiffness; Cotinine

STUDY DESIGN:
Intervention Model Description: In this prospective cohort study, women at high risk of developing preeclampsia were recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- previous smokers (Other): All women at high risk for developing preeclampsia were divided into two groups based on reported smoking status: previous smokers who quit by the positive pregnancy test, and non-smokers.
  Interventions: Other: This high-risk cohort underwent the same measurements during pregnancy: endothelial function, arterial stiffness, retinal microvasculature profile, measurement of Neprilysin, cotinine, telomere length
- non smokers (Other): All women at high risk for developing preeclampsia were divided into two groups based on reported smoking status: previous smokers who quit by the positive pregnancy test, and non-smokers.
  Interventions: Other: This high-risk cohort underwent the same measurements during pregnancy: endothelial function, arterial stiffness, retinal microvasculature profile, measurement of Neprilysin, cotinine, telomere length

INTERVENTIONS:
Other: This high-risk cohort underwent the same measurements during pregnancy: endothelial function, arterial stiffness, retinal microvasculature profile, measurement of Neprilysin, cotinine, telomere length — This high-risk cohort underwent the same measurements during pregnancy: endothelial function, arterial stiffness, retinal microvasculature profile, measurement of Neprilysin, cotinine, telomere length, and routine laboratory parameters.

SUMMARY:
This prospective cohort study explores the long-term impact of pre-pregnancy smoking on vascular health in women predisposed to preeclampsia, conducted at the Medical University of Graz. The study specifically targets women at high risk for preeclampsia who are taking aspirin as a preventative measure.

The main question it aims to answer is:

Does smoking before pregnancy influence the development and severity of preeclampsia and its associated vascular changes in high-risk women?

Participants, divided into former smokers and non-smokers, underwent comprehensive assessments throughout their pregnancies. Measurements included hemodynamic parameters such as heart rate and blood pressure, assessed with an upper arm cuff, and arterial stiffness, evaluated using pulse wave velocity with the Vicorder device. Retinal microvasculature was examined through digital imaging, and the vascular health marker ADMA, nicotine exposure marker cotinine, blood pressure regulatory enzyme neprilysin, and cellular aging indicator telomere length were quantified from blood samples. Cortisol levels were also measured from hair samples to assess stress responses.

DETAILED DESCRIPTION:
The investigators collected extensive data on each participant, including age, BMI (body mass index), and medical history, to understand their baseline health. Routine laboratory tests were conducted to monitor the health status throughout the pregnancy. Preeclampsia biomarkers and Doppler ultrasound examinations of the uterine and umbilical arteries to assess fetal and placental blood flow were conducted. The investigators tracked the development of preeclampsia, gestational hypertension (GH), and gestational diabetes mellitus (GDM).

Outcomes for the babies, such as birth weight, delivery method, gender, and the gestational week at delivery, were meticulously recorded to evaluate the broader impacts of maternal smoking and vascular health on neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

* a positive preeclampsia screening or a history of preeclampsia, daily intake of 150mg aspirin , and age over 18 years

Exclusion Criteria:

* twin pregnancies, fetal anomalies, maternal chronic renal diseases and discontinued aspirin intake.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant women at high risk for preeclampsia
Enrollment: 40 (Actual)
Dates: Start 2019-11-02 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-12-17 (Actual)

PRIMARY OUTCOMES:
Change of Pulse wave velocity | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Pulse Wave Velocity (PWV): A measure of how fast the blood pressure pulse travels through the arteries, used to assess arterial stiffness. Higher PWV indicates stiffer arteries, linked to increased cardiovascular risk.

SECONDARY OUTCOMES:
Change of Endothelial function | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Endothelial Function Assessed through ADMA: Measurement of asymmetric dimethylarginine (ADMA), an inhibitor of nitric oxide production, provides insights into endothelial health and its capacity to regulate vascular function.
Change of retinal microvasculature profile | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Retinal Microvasculature Profile Assessed through CRAE and CRVE: Central retinal arteriolar equivalent (CRAE) and central retinal venular equivalent (CRVE) are used to gauge the caliber of retinal blood vessels, reflecting systemic microvascular health.
Change of Neprilysin level | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Neprilysin levels are analyzed to understand its role in modulating vasoactive peptides, which affect blood pressure and fluid balance.
Change of Cotinine level | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Measured to determine exposure to nicotine, providing a reliable indicator of smoking status or secondhand smoke exposure.
Change of Telomere length | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Telomere Length: The measurement of telomere length serves as a biomarker of cellular aging and an indicator of potential health risks and longevity.
Blood parameters for high-risk pregnancy monitor | Measurements were conducted at three stages of pregnancy: (V1: 11-16 weeks), second trimester (V2: 24-28 weeks), and third trimester (V3: 34-37 weeks).
  Blood parameters for high-risk pregnancy monitor kidney, liver, inflammation, blood count, electrolytes, enzymes, coagulation, proteins, and placental function. Kidney: Creatinine, urea, uric acid, eGFR. Liver: Bilirubin, GGT, AST, ALT. Inflammation: CRP. Blood count: Leukocytes, erythrocytes, hemoglobin, hematocrit, MCV, MCH, MCHC, platelets, MPV. Electrolytes: Na, K, Cl, Ca, Mg. Enzymes: CK, LDH, glucose. Coagulation: PT, INR, aPTT, fibrinogen, antithrombin. Proteins: Total protein, albumin. Placental markers: sFlt-1, PlGF. These help assess maternal-fetal health, detect conditions like preeclampsia, gestational diabetes, and monitor complications in high-risk pregnancies.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided